CLINICAL TRIAL: NCT04745234
Title: Open-Label, Phase 2 Study to Assess the Safety of Mogamulizumab Given Every 4 Weeks Following Induction in Participants With Relapsed/Refractory Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: Mogamulizumab Q4week Dosing in Participants With R/R CTCL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0761-016
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Cutaneous T-Cell Lymphoma, Relapsed; Cutaneous T-Cell Lymphoma Refractory
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Recurrence | interventions — mogamulizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mogamulizumab (Experimental)
  Interventions: Drug: Mogamulizumab

INTERVENTIONS:
Drug: Mogamulizumab — For the first 28-day induction cycle (C1), mogamulizumab 1 mg/kg will be administered as an IV infusion through a 0.22- or 0.2-μm in-line filter over at least 60 minutes on Days 1, 8, 15, and 22.
  For all subsequent 28-day cycles (C2, 3, 4, etc.), mogamulizumab 2 mg/kg will be administered as an IV infusion over at least 60 minutes on Day 1 of each subsequent therapy cycle.
  Other Names: 0761, KW0761, Poteligeo

SUMMARY:
This is an open-label, multicenter, Phase 2 study to evaluate the safety and tolerability of mogamulizumab given Q4W following initial weekly induction in adult participants with relapsed/refractory MF and SS subtypes of CTCL. The study is composed of a 28-day Screening Period during which participants are screened for entry into this study, followed by a treatment period of up to 2 years from Cycle 1 Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of MF or SS

  * Stage IB, II-A, II-B, III, or IV;
* Participants who have failed at least one prior course of systemic therapy (e.g., interferon, bexarotene, photopheresis, anti-neoplastic chemotherapy). Psoralen plus ultraviolet light therapy (PUVA) is not considered a systemic therapy.

Exclusion Criteria:

* Current evidence of large cell transformation;
* Prior treatment with mogamulizumab;
* History of allogeneic transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number, percentage and severity of treatment emergent adverse events | From date of consent, at every treatment and follow up visit, up to 27 months
  Adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) (v. 5.0).

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - City of Hope National Medical Center, Duarte, California
  - University of California Irvine, Irvine, California
  - Stanford Cancer Center, Stanford, California
  - Tulane University School of Medicine, New Orleans, Louisiana
  - New York Presbyterian Hospital, New York, New York
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Hôpital Saint Louis, Paris, France
- Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Italy
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario De Salamanca, Salamanca
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No